CLINICAL TRIAL: NCT04325789
Title: A Prospective Randomized Multicenter Evaluation of Rotator Cuff Healing Using a Nanofiber Scaffold in Patients Greater Than 55 Years
Brief Title: Rotator Cuff Healing Using a Nanofiber Scaffold in Patients Greater Than 55 Years
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atreon Orthopedics (Industry)
Responsible Party: Sponsor
Organization: Nanofiber Solutions (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AO20200427
Record Dates: First submitted 2020-03-21; First posted 2020-03-30 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Tears; Full-thickness Rotator Cuff Tears
Keywords: healing; regenerative medicine; interpositional matrix; synthetic scaffold; full-thickness rotator cuff tear; enthesis regeneration
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Use of the nanofiber scaffold, in addition to SOC, during the rotator cuff repair is the intervention in this study. Study participants will be randomized into either the treatment or the control group. The control group will undergo routine rotator cuff repair without the scaffold to determine if improved healing is demonstrated with the graft.
  Group 1 (control) Group 2 (nanofiber scaffold)
Who Masked: Participant
Masking Description: This is a single blinded study. The patient will be blinded to the treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 Control (No Intervention): Group 1 will serve as the control and undergo routine rotator cuff repair with suture anchors without the nanofiber scaffold.
- Group 2 Scaffold (Active Comparator): Group 2 will undergo rotator cuff repair with suture anchors and incorporation of the nanofiber scaffold.
  Interventions: Device: nanofiber scaffold

INTERVENTIONS:
Device: nanofiber scaffold — Utilization of the interpositional nanofiber scaffold to augment the rotator cuff repair.
  Other Names: ROTIUM™ Bioresorbable Wick (Atreon Orthopedics)
  Arms: Group 2 Scaffold

SUMMARY:
Randomized controlled trial of patients over the age of 55 treated with and without a nanofiber scaffold during rotator cuff repair.

DETAILED DESCRIPTION:
1. INTRODUCTION

   This document is a protocol for a human research study. This study is to be conducted according to United States standards of Good Clinical Practice in accordance with applicable Federal regulations and institutional research policies and procedures.

   Despite numerous advancements in surgical techniques and over 250,000 procedures currently performed annually in the United States, failure of tendon healing following rotator cuff surgery occurs frequently with reports as high as 94%. Nonhealing can lead to persistent pain, poor outcomes, and a significant economic burden to society when revision surgery is required. Several factors have been associated with poor tendon healing with age greater than 60 years shown to be a significant risk factor due to diminishing vascularity at the bone tendon interface where the tear typically originates. While numerous techniques have been devised to improve fixation over the past several decades, very few have been developed to address or enhance the biology at the repair site. Rotium nanofiber is a recent FDA approved scaffold (FDA 510(K) #K183236) that has been shown to improve tendon healing to bone in animal studies. It works to mimic the extracellular matrix and helps concentrates and bind cells at the repair site providing a better organizational structure of the healing tissue. The purpose of the current study is to assess if use of the scaffold significantly improves rotator cuff healing and enhances strength in patients at higher risk of perioperative failure of the repair.
2. BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE

   Rotator cuff tears are a frequent cause of shoulder pain and disability in the elderly population. Typically, when conservative measures fail, surgery is often advised. A successful clinical outcome is felt to be heavily predicated on healing of the tendon to the bone. Despite numerous surgical and technical advancements over the past two decades not all repairs heal, with re-tear, or failure-to-heal, remaining the number one complication associated with rotator cuff surgery. This in turn creates a hefty economic burden on society whereupon surgeries are being performed with poor eventual outcomes and ultimately wasted resources.

   While reasons for failure are multifactorial, a strong correlation has been associated with advancing age. In an observational study on the natural history of rotator cuff disease, patients younger than 50 years old rarely had rotator cuff tears whereas those greater than 60 had a statistically significant greater incidence of unilateral and bilateral tears. Advancing age is believed to alter and change the intrinsic properties of the tendon leading to stiffness, hypovascularity and overall impairment of the biology of tendon healing. Furthermore, when repairs fail, they typically do so within the first four months of surgery. Means, therefore, to enhance the zone of the repair by increasing the cellularity immediately following surgery may improve the overall healing and lessen failures.

   Recently, nanofiber scaffolds have demonstrated the ability to mimic the extracellular matrix and help structure, organize, and proliferate cellular material. They do so by working, in essence, like a sponge when incorporated into the repair site, helping to bind, organize, and promote cell migration. This in effect, creates a less haphazard arrangement and induces better organization of healing tissue at the cellular level. Rotium, is an FDA-approved, nonwoven, microfiber matrix composed of PLCL (poly L-lactide-co-caprolactone) and PGL (polyglycolide) that is indicated for use in rotator cuff repair to enhance healing at the bone tendon interface. The implant is inserted under the rotator cuff tendon and placed on top of the greater tuberosity at the time of surgery and typically positioned over a suture. In a recent animal study performed at Colorado State University, a nearly 75% increased strength of repair was demonstrated at twelve weeks in those tendons treated with the graft. This will be the first prospective randomized clinical study in humans assessing for a difference in healing and strength in a population of patients considered at high risk for postoperative failure of the repair.
3. STUDY OBJECTIVES

Utilizing a randomized controlled trial, this study seeks to evaluate if there is a difference in post-operative healing, strength, and functional outcomes in patients older than 55 years with rotator cuff tears treated with and without the nanofiber scaffold.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55 and older
2. Able to provide informed consent
3. Primary diagnosis of rotator cuff tear

Exclusion Criteria:

1. Revision rotator cuff surgery
2. Partial thickness rotator cuff tears
3. Massive (greater than 5cm) rotator cuff tears
4. Patients with current tobacco history

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Failure of the repair | 24 months
  To determine if the use of the nanofiber scaffold changes the occurrence of postoperative rotator cuff repair (RCR) failure in patients older than 55 years

SECONDARY OUTCOMES:
Change in shoulder range of motion | Preoperative, 6 weeks, 3 months, 6 months, 12 months, 24 months postoperative
  Patients range of motion including forward flexion, abduction and external rotation will be measured preopertively and postoperatively with a manual goniometer at 6 weeks, 3 months, 6 months, 12 months and 24 months postoperatively to measure for differences.
Change in isometric rotator cuff muscle strength peak force | Preoperative, 3 months, 6 months, 12 months, 24 months postoperative
  To determine if the use of the nanofiber scaffold changes postoperative isometric muscle strength following RCR using a Lafayette muscle dynometer. The contralateral shoulder will be assessed for comparison. Measurements will be recorded in peak force and pounds of force.
Change in patient-reported American Shoulder and Elbow Scores | Preoperative, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months postoperative
  To determine if there is a difference in American Shoulder and Elbow scores of patients with rotator cuff tears treated with and without the nanofiber scaffold measured at preoperative visit, 2 weeks, 6 weeks, 3 months, 6 months, 12 months and 24 months after surgery.
Change in patient-reported postoperative pain (Visual Analogue Scale - Pain) | Preoperative, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months postoperative
  Patient reported postoperative visual analogue pain (on a scale of 0-10), measured preoperatively and postoperatively will be assessed for a difference. Pain scores will be checked at 2 weeks, 6 weeks, 3 months, 6 months, 12 months and 24 months after surgery.
Change in patient-reported Single Assessment Numeric Evaluation (SANE) score | Preoperative, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months postoperative
  Patient reported SANE score (on a scale of 0 to 100%), measured preoperatively and postoperatively will be assessed for a difference; Scores will be checked at 2 weeks, 6 weeks, 3 months, 6 months, 12 months and 24 months after surgery.
Change in patient-reported Veteran Rand 12 (VR-12) score | Preoperative, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months postoperative
  Patient reported VR-12 (Veteran rand) will be compared measured postoperatively will be assessed for a difference; Scores will be checked at 2 weeks, 6 weeks, 3 months, 6 months, 12 months and 24 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Badman, MD, Principal Investigator — Central Indiana Orthopedics; Elsa I Englund Kayuha, MD, Study Director — Atreon Orthopedics
Locations (4):
- United States (4):
  - Central Indiana Orthopedics, Fishers, Indiana
  - Associated Orthopedists of Detroit, Saint Clair Shores, Michigan
  - The Christ Hospital & The Lindner Reseach Center at The Christ Hospital, Cincinnati, Ohio
  - Steadman Hawkins Clinic of the Carolinas - Patewood, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mather RC 3rd, Koenig L, Acevedo D, Dall TM, Gallo P, Romeo A, Tongue J, Williams G Jr. The societal and economic value of rotator cuff repair. J Bone Joint Surg Am. 2013 Nov 20;95(22):1993-2000. doi: 10.2106/JBJS.L.01495. PMID 24257656
- [Background] Harryman DT 2nd, Hettrich CM, Smith KL, Campbell B, Sidles JA, Matsen FA 3rd. A prospective multipractice investigation of patients with full-thickness rotator cuff tears: the importance of comorbidities, practice, and other covariables on self-assessed shoulder function and health status. J Bone Joint Surg Am. 2003 Apr;85(4):690-6. PMID 12672846
- [Background] Iannotti JP, Deutsch A, Green A, Rudicel S, Christensen J, Marraffino S, Rodeo S. Time to failure after rotator cuff repair: a prospective imaging study. J Bone Joint Surg Am. 2013 Jun 5;95(11):965-71. doi: 10.2106/JBJS.L.00708. PMID 23780533
- [Background] Agudelo-Garcia PA, De Jesus JK, Williams SP, Nowicki MO, Chiocca EA, Liyanarachchi S, Li PK, Lannutti JJ, Johnson JK, Lawler SE, Viapiano MS. Glioma cell migration on three-dimensional nanofiber scaffolds is regulated by substrate topography and abolished by inhibition of STAT3 signaling. Neoplasia. 2011 Sep;13(9):831-40. doi: 10.1593/neo.11612. PMID 21969816
- [Background] Teunis T, Lubberts B, Reilly BT, Ring D. A systematic review and pooled analysis of the prevalence of rotator cuff disease with increasing age. J Shoulder Elbow Surg. 2014 Dec;23(12):1913-1921. doi: 10.1016/j.jse.2014.08.001. PMID 25441568
- [Background] Le BT, Wu XL, Lam PH, Murrell GA. Factors predicting rotator cuff retears: an analysis of 1000 consecutive rotator cuff repairs. Am J Sports Med. 2014 May;42(5):1134-42. doi: 10.1177/0363546514525336. Epub 2014 Apr 18. PMID 24748610
- [Background] Diebold G, Lam P, Walton J, Murrell GAC. Relationship Between Age and Rotator Cuff Retear: A Study of 1,600 Consecutive Rotator Cuff Repairs. J Bone Joint Surg Am. 2017 Jul 19;99(14):1198-1205. doi: 10.2106/JBJS.16.00770. PMID 28719559
- [Background] Gulotta LV, Nho SJ, Dodson CC, Adler RS, Altchek DW, MacGillivray JD; HSS Arthroscopic Rotator Cuff Registry. Prospective evaluation of arthroscopic rotator cuff repairs at 5 years: part II--prognostic factors for clinical and radiographic outcomes. J Shoulder Elbow Surg. 2011 Sep;20(6):941-6. doi: 10.1016/j.jse.2011.03.028. Epub 2011 Jun 29. PMID 21719319
- [Background] Liem D, Lichtenberg S, Magosch P, Habermeyer P. Magnetic resonance imaging of arthroscopic supraspinatus tendon repair. J Bone Joint Surg Am. 2007 Aug;89(8):1770-6. doi: 10.2106/JBJS.F.00749. PMID 17671017
- [Background] Koh KH, Kang KC, Lim TK, Shon MS, Yoo JC. Prospective randomized clinical trial of single- versus double-row suture anchor repair in 2- to 4-cm rotator cuff tears: clinical and magnetic resonance imaging results. Arthroscopy. 2011 Apr;27(4):453-62. doi: 10.1016/j.arthro.2010.11.059. PMID 21444007
- [Background] Boileau P, Brassart N, Watkinson DJ, Carles M, Hatzidakis AM, Krishnan SG. Arthroscopic repair of full-thickness tears of the supraspinatus: does the tendon really heal? J Bone Joint Surg Am. 2005 Jun;87(6):1229-40. doi: 10.2106/JBJS.D.02035. PMID 15930531
- [Background] Tempelhof S, Rupp S, Seil R. Age-related prevalence of rotator cuff tears in asymptomatic shoulders. J Shoulder Elbow Surg. 1999 Jul-Aug;8(4):296-9. doi: 10.1016/s1058-2746(99)90148-9. PMID 10471998
- [Background] Bishop J, Klepps S, Lo IK, Bird J, Gladstone JN, Flatow EL. Cuff integrity after arthroscopic versus open rotator cuff repair: a prospective study. J Shoulder Elbow Surg. 2006 May-Jun;15(3):290-9. doi: 10.1016/j.jse.2005.09.017. PMID 16679227
- [Background] Tashjian RZ, Hollins AM, Kim HM, Teefey SA, Middleton WD, Steger-May K, Galatz LM, Yamaguchi K. Factors affecting healing rates after arthroscopic double-row rotator cuff repair. Am J Sports Med. 2010 Dec;38(12):2435-42. doi: 10.1177/0363546510382835. Epub 2010 Oct 28. PMID 21030564
- [Background] Thomazeau H, Boukobza E, Morcet N, Chaperon J, Langlais F. Prediction of rotator cuff repair results by magnetic resonance imaging. Clin Orthop Relat Res. 1997 Nov;(344):275-83. PMID 9372778
- [Background] Kim KC, Shin HD, Lee WY. Repair integrity and functional outcomes after arthroscopic suture-bridge rotator cuff repair. J Bone Joint Surg Am. 2012 Apr 18;94(8):e48. doi: 10.2106/JBJS.K.00158. PMID 22517394
- [Background] Boehm TD, Werner A, Radtke S, Mueller T, Kirschner S, Gohlke F. The effect of suture materials and techniques on the outcome of repair of the rotator cuff: a prospective, randomised study. J Bone Joint Surg Br. 2005 Jun;87(6):819-23. doi: 10.1302/0301-620X.87B6.15638. PMID 15911666
- [Background] Charousset C, Grimberg J, Duranthon LD, Bellaiche L, Petrover D. Can a double-row anchorage technique improve tendon healing in arthroscopic rotator cuff repair?: A prospective, nonrandomized, comparative study of double-row and single-row anchorage techniques with computed tomographic arthrography tendon healing assessment. Am J Sports Med. 2007 Aug;35(8):1247-53. doi: 10.1177/0363546507301661. Epub 2007 Apr 23. PMID 17452513
- [Background] Deutsch A, Kroll DG, Hasapes J, Staewen RS, Pham C, Tait C. Repair integrity and clinical outcome after arthroscopic rotator cuff repair using single-row anchor fixation: a prospective study of single-tendon and two-tendon tears. J Shoulder Elbow Surg. 2008 Nov-Dec;17(6):845-52. doi: 10.1016/j.jse.2008.04.004. Epub 2008 Aug 20. PMID 18718766
- [Background] Franceschi F, Ruzzini L, Longo UG, Martina FM, Zobel BB, Maffulli N, Denaro V. Equivalent clinical results of arthroscopic single-row and double-row suture anchor repair for rotator cuff tears: a randomized controlled trial. Am J Sports Med. 2007 Aug;35(8):1254-60. doi: 10.1177/0363546507302218. Epub 2007 Jun 6. PMID 17554104
- [Background] Klepps S, Bishop J, Lin J, Cahlon O, Strauss A, Hayes P, Flatow EL. Prospective evaluation of the effect of rotator cuff integrity on the outcome of open rotator cuff repairs. Am J Sports Med. 2004 Oct-Nov;32(7):1716-22. doi: 10.1177/0363546504265262. PMID 15494338
- [Background] Ko SH, Lee CC, Friedman D, Park KB, Warner JJ. Arthroscopic single-row supraspinatus tendon repair with a modified mattress locking stitch: a prospective, randomized controlled comparison with a simple stitch. Arthroscopy. 2008 Sep;24(9):1005-12. doi: 10.1016/j.arthro.2008.04.074. Epub 2008 Jun 24. PMID 18760207
- [Background] Lapner PL, Sabri E, Rakhra K, McRae S, Leiter J, Bell K, Macdonald P. A multicenter randomized controlled trial comparing single-row with double-row fixation in arthroscopic rotator cuff repair. J Bone Joint Surg Am. 2012 Jul 18;94(14):1249-57. doi: 10.2106/JBJS.K.00999. PMID 22810395
- [Background] Lee BG, Cho NS, Rhee YG. Effect of two rehabilitation protocols on range of motion and healing rates after arthroscopic rotator cuff repair: aggressive versus limited early passive exercises. Arthroscopy. 2012 Jan;28(1):34-42. doi: 10.1016/j.arthro.2011.07.012. Epub 2011 Oct 20. PMID 22014477
- [Background] Ma HL, Chiang ER, Wu HT, Hung SC, Wang ST, Liu CL, Chen TH. Clinical outcome and imaging of arthroscopic single-row and double-row rotator cuff repair: a prospective randomized trial. Arthroscopy. 2012 Jan;28(1):16-24. doi: 10.1016/j.arthro.2011.07.003. Epub 2011 Oct 7. PMID 21982391
- [Background] Galatz LM, Ball CM, Teefey SA, Middleton WD, Yamaguchi K. The outcome and repair integrity of completely arthroscopically repaired large and massive rotator cuff tears. J Bone Joint Surg Am. 2004 Feb;86(2):219-24. doi: 10.2106/00004623-200402000-00002. PMID 14960664
- [Background] Jost B, Pfirrmann CW, Gerber C, Switzerland Z. Clinical outcome after structural failure of rotator cuff repairs. J Bone Joint Surg Am. 2000 Mar;82(3):304-14. doi: 10.2106/00004623-200003000-00002. PMID 10724223
- [Background] Liu SH, Baker CL. Arthroscopically assisted rotator cuff repair: correlation of functional results with integrity of the cuff. Arthroscopy. 1994 Feb;10(1):54-60. doi: 10.1016/s0749-8063(05)80293-2. PMID 8166903
- [Background] Akpinar S, Uysal M, Pourbagher MA, Ozalay M, Cesur N, Hersekli MA. Prospective evaluation of the functional and anatomical results of arthroscopic repair in small and medium-sized full-thickness tears of the supraspinatus tendon. Acta Orthop Traumatol Turc. 2011;45(4):248-53. doi: 10.3944/AOTT.2011.2455. PMID 21908964
- [Background] Harryman DT 2nd, Mack LA, Wang KY, Jackins SE, Richardson ML, Matsen FA 3rd. Repairs of the rotator cuff. Correlation of functional results with integrity of the cuff. J Bone Joint Surg Am. 1991 Aug;73(7):982-9. PMID 1874784
- [Background] Mall NA, Kim HM, Keener JD, Steger-May K, Teefey SA, Middleton WD, Stobbs G, Yamaguchi K. Symptomatic progression of asymptomatic rotator cuff tears: a prospective study of clinical and sonographic variables. J Bone Joint Surg Am. 2010 Nov 17;92(16):2623-33. doi: 10.2106/JBJS.I.00506. PMID 21084574
- [Background] Yamaguchi K, Ditsios K, Middleton WD, Hildebolt CF, Galatz LM, Teefey SA. The demographic and morphological features of rotator cuff disease. A comparison of asymptomatic and symptomatic shoulders. J Bone Joint Surg Am. 2006 Aug;88(8):1699-704. doi: 10.2106/JBJS.E.00835. PMID 16882890
- [Background] Cho NS, Rhee YG. The factors affecting the clinical outcome and integrity of arthroscopically repaired rotator cuff tears of the shoulder. Clin Orthop Surg. 2009 Jun;1(2):96-104. doi: 10.4055/cios.2009.1.2.96. Epub 2009 May 30. PMID 19885061
- [Background] Nho SJ, Shindle MK, Adler RS, Warren RF, Altchek DW, MacGillivray JD. Prospective analysis of arthroscopic rotator cuff repair: subgroup analysis. J Shoulder Elbow Surg. 2009 Sep-Oct;18(5):697-704. doi: 10.1016/j.jse.2008.11.018. Epub 2009 Mar 9. PMID 19269861
- [Background] Hein J, Reilly JM, Chae J, Maerz T, Anderson K. Retear Rates After Arthroscopic Single-Row, Double-Row, and Suture Bridge Rotator Cuff Repair at a Minimum of 1 Year of Imaging Follow-up: A Systematic Review. Arthroscopy. 2015 Nov;31(11):2274-81. doi: 10.1016/j.arthro.2015.06.004. Epub 2015 Jul 15. PMID 26188783
- [Background] Fukunishi T, Best CA, Ong CS, Groehl T, Reinhardt J, Yi T, Miyachi H, Zhang H, Shinoka T, Breuer CK, Johnson J, Hibino N. Role of Bone Marrow Mononuclear Cell Seeding for Nanofiber Vascular Grafts. Tissue Eng Part A. 2018 Jan;24(1-2):135-144. doi: 10.1089/ten.TEA.2017.0044. Epub 2017 Jun 13. PMID 28486019
- [Background] Fukunishi T, Best CA, Sugiura T, Opfermann J, Ong CS, Shinoka T, Breuer CK, Krieger A, Johnson J, Hibino N. Preclinical study of patient-specific cell-free nanofiber tissue-engineered vascular grafts using 3-dimensional printing in a sheep model. J Thorac Cardiovasc Surg. 2017 Apr;153(4):924-932. doi: 10.1016/j.jtcvs.2016.10.066. Epub 2016 Nov 14. PMID 27938900
- [Background] Romeo A, Easley J, Regan D, Hackett E, Johnson J, Johnson J, Puttlitz C, McGilvray K. Rotator cuff repair using a bioresorbable nanofiber interposition scaffold: a biomechanical and histologic analysis in sheep. J Shoulder Elbow Surg. 2022 Feb;31(2):402-412. doi: 10.1016/j.jse.2021.07.018. Epub 2021 Aug 25. PMID 34454041